CLINICAL TRIAL: NCT03347721
Title: Does Lidocaine Gel Decrease Pain Perception in Women Undergoing Diagnostic Flexible Cystoscopy?
Brief Title: Does Lidocaine Gel Decrease Pain Perception in Women Undergoing Diagnostic Flexible Cystoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Erin Dougher, Principal Investigator, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 9504
Record Dates: First submitted 2017-11-13; First posted 2017-11-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Cystoscopy; Lidocaine; Pain Perception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine gel (Active Comparator)
  Interventions: Drug: lidocaine gel
- Lubricant Gel (Placebo Comparator)
  Interventions: Drug: Lubricant Gel

INTERVENTIONS:
Drug: lidocaine gel — 2% lidocaine jelly, injected into the urethra
  Arms: Lidocaine gel
Drug: Lubricant Gel — Lubricating gel
  Other Names: Plain gel
  Arms: Lubricant Gel

SUMMARY:
This study is to determine if there is a clinically meaningful difference in pain perception for women during in-office diagnostic flexible cystoscopy when using lidocaine gel vs plain lubricant. This will be a double blinded randomized control trial.

DETAILED DESCRIPTION:
The use of anesthetic lubricant during in-office flexible cystoscopy has been well studied men. Pain during cystoscopy can lead to poor compliance and follow-up. Very few studies challenging the use of anesthetic lubricant during cystoscopy have included women. Those that have, only recruited a small number with insignificant findings. A meta-analysis reviewed four studies looking at the efficacy of lidocaine gel on pain relief during flexible cystoscopy in men. Four hundred and eleven men underwent flexible cystoscopy with and without the use of lidocaine gel and those who received anesthetic gel were 1.7 times more likely not to experience moderate to severe pain than those who received placebo. The anatomy of the female and male urogenital tract differ. The female urethra is approximately 3cm in length while the male urethra averages 7 cm with an external and prostatic sphincter which is the location where the most discomfort is thought to occur. A randomized control trial of 144 women undergoing rigid cystoscopy and found that pain was decreased with lidocaine vs placebo, however other studies such found no difference in pain perception. The efficacy of lidocaine gel in women during flexible cystoscopy has not been studied. The use of lidocaine gel during diagnostic flexible cystoscopy in women is based on surgeon preference and experience, and use of either plain or anesthetic gel, is currently acceptable clinical practice. The morbidity and cost of local anesthesia associated with cystoscopy in women is unknown due to the lack of studies. The objective of this study is to determine if there is a clinically meaningful difference in pain perception in women during in-office diagnostic flexible cystoscopy when using lidocaine gel vs plain lubricant.

ELIGIBILITY:
Inclusion Criteria:

* need for in office diagnostic flexible cystoscopy

Exclusion Criteria:

* urethral stricture
* simultaneous scheduling or performed additional procedure
* current urinary tract infection
* hypersensitivity to local anesthetic of amide type

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain and satisfaction | Recorded immediately after the procedure
  Composite of pain and satisfaction as determined by a Numeric Rating Scale for pain (validated measure) rating pain, as well as answers to yes or no questions asking if patient would repeat procedure in same method and if pain medicine is needed at end of procedure.

SECONDARY OUTCOMES:
Anticipated pain | Recorded prior to procedure at time of enrollment into study (anticipated) and immediately after procedure
  Composite of pain anticipated during procedure and compared to actual pain perceived as determined by a Numeric Rating Scale for pain (validated measure) rating pain

CONTACTS AND LOCATIONS:
Locations (1):
- Louisiana State University- Health Science Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No